CLINICAL TRIAL: NCT07020052
Title: Phase II Exploratory Study of Sequential Triple Therapy (Temozolomide/Anlotinib/Bemarituzumab) in Combination With Concurrent Radiotherapy With Temozolomide and Anlotinib for the Maintenance Treatment of Diffuse Midline Gliomas in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, kunyu yang, Director of Oncology Department, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: DMGtriple2025
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Maintenance Treatment of Diffuse Midline Gliomas in Children
MeSH Terms: interventions — Temozolomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples were collected from all subjects in this study for blood routine, biochemical, cellular subpopulation, and cytokine testing at each visit (M3, M6, M9, M12) during the infusion period (D0), treatment period, and follow-up period. The results of cytokines during this stage will be used as an indicator for pharmacodynamic (PD) evaluation. The relevant testing is completed by the Inspection Department of our hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- triple therapy: Starting from 30 days after radiotherapy, adjuvant temozolomide was orally administered at a dose of 150mg/m2. The dosage of temozolomide was adjusted to 200mg/m2 starting from the second cycle, with continuous use for 5 days per week and a 23 day hiatus. Oral administration for a total of 6 cycles.
  The start time of oral administration of anlotinib after radiotherapy follows the cycle of radiotherapy, with continuous oral administration for 2 weeks and cessation for 1 week. Until the side effects are intolerable or the tumor progresses. The maximum duration shall not exceed 24 months.
  Begin treatment with bemarituzumab 24 hours after radiotherapy, with a body weight of>=45kg, intravenous injection of 200mg, once every 3 weeks. Weight<45kg, 100mg intravenous injection, once every 3 weeks. Until the side effects are intolerable or the tumor progresses. The maximum duration shall not exceed 24 months.
  Interventions: Drug: temozolomide/anlotinib/pembrolizumab

INTERVENTIONS:
Drug: temozolomide/anlotinib/pembrolizumab — Starting from 30 days after radiotherapy, adjuvant temozolomide was orally administered at a dose of 150mg/m2. The dosage of temozolomide was adjusted to 200mg/m2 starting from the second cycle, with continuous use for 5 days per week and a 23 day hiatus. Oral administration for a total of 6 cycles.
  The start time of oral administration of anlotinib after radiotherapy follows the cycle of radiotherapy, with continuous oral administration for 2 weeks and cessation for 1 week. Until the side effects are intolerable or the tumor progresses. The maximum duration shall not exceed 24 months.
  Begin treatment with bemarituzumab 24 hours after radiotherapy, with a body weight of>=45kg, intravenous injection of 200mg, once every 3 weeks. Weight<45kg, 100mg intravenous injection, once every 3 weeks. Until the side effects are intolerable or the tumor progresses. The maximum duration shall not exceed 24 months.

SUMMARY:
This study is a phase II single center exploratory clinical trial aimed at evaluating the efficacy and safety of temozolomide combined with anlotinib synchronous radiotherapy sequential triple therapy (temozolomide/anlotinib/PD-L1 inhibitor) for the maintenance treatment of diffuse midline gliomas (DMG) in children. The research plan includes 33 children with DMG aged 3-18 years, who have been pathologically diagnosed and have not received systematic treatment. The implementation will be divided into two stages: synchronous radiotherapy and chemotherapy stage (54Gy radiotherapy+oral temozolomide 75mg/m ²+sequential oral anlotinib) and maintenance treatment stage (increasing temozolomide dose+continuous use of anlotinib+intravenous injection of PD-L1 inhibitor according to body weight). Through multi mechanism synergy (radiotherapy sensitization, anti angiogenesis, and immune activation), the limitations of traditional treatment will be overcome. The primary endpoint is progression free survival (PFS), while secondary endpoints include objective response rate (ORR), 2-year overall survival rate (2y OS), quality of life, and safety (CTCAE 4.0 criteria). The innovation of the research lies in the first proposal of a "synchronous maintenance" staged mode, targeting the molecular characteristics of DMG (H3K27M mutation), combined with previous evidence at home and abroad (such as the median PFS of 10.2 months for anlotinib combined with synchronous radiotherapy), aiming to provide a new comprehensive treatment plan for this highly invasive tumor.

ELIGIBILITY:
inclusion criteria 1.Age 3-18 years old, gender not limited； 2. Pathological diagnosis of diffuse midline gliomas in children;； 3. Not achieving complete surgical resection； 4. According to the 2021 WHO Classification of Central Nervous System Tumors (Fifth Edition) ； 5. Have not received specialized treatment for diffuse midline gliomas in children in the past;； 6. According to RECIST version 1.1 standard, at least one assessable target lesion is required; 7. ECOG physical fitness status is 0-4 points; 8. The main organ function is normal, which meets the following criteria:

1. The standard for blood routine examination must meet the following criteria: (no blood transfusion within 14 days)

   1. Hb≥90g/L:
   2. ANC≥1.5*10^9/L;
   3. PLT≥80*10^9／L；
2. Biochemical tests must meet the following standards

   1. BIL<1.25 times the upper limit of normal (ULN);
   2. ALT and AST<2.5*ULN;
   3. Serum Cr ≤ ULN, endogenous creatinine clearance rate>50ml/min (Cockcroft Gaut formula); 9. Sign a written informed consent form before conducting any experimental activities; 10. Researchers determine that they are able to comply with the research protocol; 11. Negative pregnancy test (for female patients with fertility) during screening; 12. Male patients with fertility and female patients with fertility and pregnancy risk must agree to use two contraceptive methods throughout the study period (at least one of which is considered an effective contraceptive method).

      Female patients who do not have fertility (i.e. meet at least one of the following criteria):
      * Have undergone hysterectomy and/or bilateral oophorectomy with documented records;
      * medically confirmed ovarian dysfunction;
      * Postmenopausal status, defined as a state of continuous cessation of menstruation for at least 12 months without other pathological or physiological reasons, and confirmed by serum follicle stimulating hormone (FSH) levels consistent with postmenopausal status.

      A signed and dated informed consent form indicating that the patient (or legal representative, if permitted by local guidelines/practices) has been informed of all relevant aspects of the study.

      13. Patients who are willing and able to comply with visit arrangements, treatment plans, laboratory tests, and other research procedures.

      exclusion criteria
      1. Previously received anti-tumor treatment for diffuse midline glioma;
      2. Previous or concurrent malignant tumors (excluding malignant tumors that have been cured and have a cancer free survival of more than 5 years, such as basal cell carcinoma of the skin, cervical carcinoma in situ, and papillary thyroid carcinoma);
      3. Uncontrolled clinical symptoms or diseases of the heart, such as: (1) NYHA grade II or above heart failure (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention in patients;
      4. Active infections that require treatment;
      5. People with congenital or acquired immune deficiency (such as HIV infected people), active hepatitis B (HBV-DNA ≥ 104 copies/ml or 2000IU/ml) or hepatitis C (hepatitis C antibody is positive, and HCV-RNA is higher than the detection limit of the analytical method);
      6. Known history of substance abuse, alcoholism, or drug use;
      7. According to the researcher's judgment, there may be other factors that could force the subject to terminate the study midway, such as suffering from other serious illnesses (including mental illnesses) that require concurrent treatment, severe abnormal laboratory test values, family or social factors that may affect the subject's safety or the collection of trial data;
      8. Patients who the surgeon believes can undergo curative resection;
      9. Active pulmonary tuberculosis;
      10. Serious infections (including but not limited to hospitalization due to infection, bacteremia, or complications of severe pneumonia) that occurred within 4 weeks prior to the start of the study treatment.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with diffuse midline glioma diagnosed by pathology.
Sampling Method: Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2030-04-10 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 5years
  The survival time of no progression in tumor after therapy

SECONDARY OUTCOMES:
ORR | 3 months
  objective relief rate
2-year OS | 2 years
  overall survival rate in 2years

CONTACTS AND LOCATIONS:
Locations (1):
- inyinhu Cancer Center, UnionMedical College Affiliated Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cohen EE, Karrison TG, Kocherginsky M, Mueller J, Egan R, Huang CH, Brockstein BE, Agulnik MB, Mittal BB, Yunus F, Samant S, Raez LE, Mehra R, Kumar P, Ondrey F, Marchand P, Braegas B, Seiwert TY, Villaflor VM, Haraf DJ, Vokes EE. Phase III randomized trial of induction chemotherapy in patients with N2 or N3 locally advanced head and neck cancer. J Clin Oncol. 2014 Sep 1;32(25):2735-43. doi: 10.1200/JCO.2013.54.6309. Epub 2014 Jul 21. PMID 25049329
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Ogino T, Shigyo H, Ishii H, Katayama A, Miyokawa N, Harabuchi Y, Ferrone S. HLA class I antigen down-regulation in primary laryngeal squamous cell carcinoma lesions as a poor prognostic marker. Cancer Res. 2006 Sep 15;66(18):9281-9. doi: 10.1158/0008-5472.CAN-06-0488. PMID 16982773
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Faivre-Finn C, Reck M, Vansteenkiste J, Spigel DR, Wadsworth C, Melillo G, Taboada M, Dennis PA, Ozguroglu M; PACIFIC Investigators. Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC. N Engl J Med. 2018 Dec 13;379(24):2342-2350. doi: 10.1056/NEJMoa1809697. Epub 2018 Sep 25. PMID 30280658
- [Background] Gandhi L, Rodriguez-Abreu D, Gadgeel S, Esteban E, Felip E, De Angelis F, Domine M, Clingan P, Hochmair MJ, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Hui R, Garon EB, Boyer M, Rubio-Viqueira B, Novello S, Kurata T, Gray JE, Vida J, Wei Z, Yang J, Raftopoulos H, Pietanza MC, Garassino MC; KEYNOTE-189 Investigators. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med. 2018 May 31;378(22):2078-2092. doi: 10.1056/NEJMoa1801005. Epub 2018 Apr 16. PMID 29658856
- [Background] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012
- [Background] Eason T, Mihalko W, Toy PC. Robotic-Assisted Total Knee Arthroplasty is Safe in the Ambulatory Surgery Center Setting. Orthop Clin North Am. 2023 Apr;54(2):153-159. doi: 10.1016/j.ocl.2022.11.001. PMID 36894288
- [Background] Wolff HA, Overbeck T, Roedel RM, Hermann RM, Herrmann MK, Kertesz T, Vorwerk H, Hille A, Matthias C, Hess CF, Christiansen H. Toxicity of daily low dose cisplatin in radiochemotherapy for locally advanced head and neck cancer. J Cancer Res Clin Oncol. 2009 Jul;135(7):961-7. doi: 10.1007/s00432-008-0532-x. Epub 2008 Dec 24. PMID 19107519
- [Background] Yu Y, Yang G, Huang H, Fu Z, Cao Z, Zheng L, You L, Zhang T. Preclinical models of pancreatic ductal adenocarcinoma: challenges and opportunities in the era of precision medicine. J Exp Clin Cancer Res. 2021 Jan 5;40(1):8. doi: 10.1186/s13046-020-01787-5. PMID 33402215